CLINICAL TRIAL: NCT04336826
Title: An Open-Label Study Evaluating the Safety and Pharmacokinetics of Ataluren in Children From ≥6 Months to <2 Years of Age With Nonsense Mutation Duchenne Muscular Dystrophy
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of Ataluren in Participants From ≥6 Months to <2 Years of Age With Nonsense Mutation Duchenne Muscular Dystrophy (nmDMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-048-DMD; 2020-000980-21 (EudraCT Number)
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-02

CONDITIONS: Nonsene Mutation Duchenne Muscular Dystrophy
MeSH Terms: interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ataluren (Experimental): Participants will receive ataluren oral suspension 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening each day for 24 weeks.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren will be administered as per the dose and schedule specified in the arm.
  Other Names: PTC124

SUMMARY:
This study is designed to evaluate safety, tolerability, and pharmacokinetics (PK) in male children with nmDMD aged ≥6 months to <2 years treated daily for 24 weeks with orally administered ataluren 10, 10, and 20 milligrams/kilogram (mg/kg) (morning, mid-day, and evening dose, respectively).

DETAILED DESCRIPTION:
Participants who complete the 24-week treatment period in this study will be offered participation to a follow-up extension period for at least 52 weeks from the date of first administration of ataluren in this parent study.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥7.5 kilograms (kg)
* Diagnosis of duchenne muscular dystrophy (DMD) based on an elevated serum creatine kinase and genotypic evidence of dystrophinopathy.
* Documentation of the presence of a nonsense mutation of the dystrophin gene as determined by gene sequencing prior to enrollment.

Exclusion Criteria:

* Participation in any drug or device investigation or whose sibling is currently participating in a blinded portion of another ataluren study or received an investigational drug within three months prior to the Screening Visit or who anticipate participating in any other drug or device clinical investigation or receiving any other investigational drug within the duration of this study.
* Expectation of a major surgical procedure during the study period.
* Known hypersensitivity to any of the ingredients or excipients of the study drug (polydextrose, polyethylene glycol 3350, poloxamer 407, mannitol 25C, crospovidone XL10, hydroxyethyl cellulose, vanilla, colloidal silica, or magnesium stearate).
* Ongoing use of the following drugs:

  1. Systemic aminoglycoside therapy and/or intravenous (IV) vancomycin.
  2. Coumarin-based anticoagulants (for example, warfarin), phenytoin, tolbutamide, or paclitaxel.
  3. Inducers of UGT1A9 (for example, rifampicin), or substrates of OAT1 or OAT3 (for example, ciprofloxacin, adefovir, oseltamivir, aciclovir, captopril, furosemide, bumetanide, valsartan, pravastatin, rosuvastatin, atorvastatin, pitavastatin).

Ages: 6 Months to 2 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Penematsa, Study Director — PTC Therapeutics, Inc.
Locations (1):
- Rare Disease Research, LLC, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ataluren: Participants received ataluren oral suspension 10 milligrams (mg)/kilogram (kg) in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening each day for up to 24 weeks.
Period: Overall Study
Arm/Group | Ataluren
Started | 6
Received at Least 1 Dose of Study Drug | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of ataluren.
Groups:
- Ataluren: Participants received ataluren oral suspension 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening each day for up to 24 weeks.
Arm/Group | Ataluren
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.153 (0.4485)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Serious adverse event (SAE): an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect, important medical event. A TEAE was defined as an AE that occurred or worsened while on ataluren (on or after first dose of ataluren) up to 4 weeks after the last dose. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to Week 28
Population: Safety analysis set included all participants who received at least 1 dose of ataluren.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 6
Participants | 5

2. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24) of Ataluren
Time Frame: Predose up to 12 hours postdose at Week 24
Population: PK population included all participants who received at least 1 dose of ataluren and had 1 PK concentration datum. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*micrograms (μg)/milliliter (mL)
Arm/Group | Ataluren
Number analyzed (Participants) | 4
hours*micrograms (μg)/milliliter (mL) | 167 (23.8)

3. Secondary Outcome: Area Under the Concentration-Time Curve Between Dosing Interval (AUC0-τ) of Ataluren
Time Frame: Predose up to 12 hours postdose at Week 24
Population: PK population included all participants who received at least 1 dose of ataluren and had 1 PK concentration datum.
Measure: Mean (Standard Deviation); unit: hours*μg/mL
Arm/Group | Ataluren
Number analyzed (Participants) | 6
hours*μg/mL | NA (NA) — Per prespecified analysis, 'Measure Type' and 'Method of Dispersion' were not estimable for this outcome measure because there were insufficient number of participants with data within the linear regression of concentration in the logarithmic scale versus time.

4. Secondary Outcome: Maximum Concentration (Cmax) of Ataluren
Time Frame: Predose up to 12 hours postdose at Week 24
Population: PK population included all participants who received at least 1 dose of ataluren and had 1 PK concentration datum.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Ataluren
Number analyzed (Participants) | 6
μg/mL | 12.6 (3.64)

5. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Ataluren
Time Frame: Predose up to 12 hours postdose at Week 24
Population: PK population included all participants who received at least 1 dose of ataluren and had 1 PK concentration datum.
Measure: Median (Full Range); unit: hours
Arm/Group | Ataluren
Number analyzed (Participants) | 6
hours | 2.08 [1.00 to 4.13]

6. Secondary Outcome: Trough Concentration (Ctrough) of Ataluren
Time Frame: Predose up to 12 hours postdose at Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Ataluren
Number analyzed (Participants) | 5
μg/mL | 3.48 (3.36)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 28
Description: Safety analysis set included all participants who received at least 1 dose of ataluren.
Arm/Group | Ataluren
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=6)
Diarrhoea (Gastrointestinal disorders) | 2
Teething (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Body tinea (Infections and infestations) | 1
Enterovirus infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Hand-foot-and-mouth disease (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Skin plaque (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT04336826/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT04336826/SAP_001.pdf